CLINICAL TRIAL: NCT00043264
Title: Antibiotic Treatment Trial Directed Against Chlamydia Pneumonia in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Multiple Sclerosis Society (Other)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR02558-0176
Record Dates: First submitted 2002-08-07; First posted 2002-08-08 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rifampin; Azithromycin

INTERVENTIONS:
Drug: Rifampin
Drug: Azithromycin

SUMMARY:
Multiple sclerosis (MS) is an inflammatory, demyelinating disease which affects the central nervous system (CNS). The etiology of MS is unknown, although the immune system appears to play a role. Many different infectious agents have been proposed as potential causes for MS, including Epstein-Barr virus, human herpesvirus 6, and coronaviruses. Recently Dr. Sriram at Vanderbilt University has found evidence for active Chlamydia pneumonia infection in the CNS of MS patients. These findings have been replicated in part by other laboratories.

The purpose of the current study is to test whether antibiotic treatment aimed at eradicating Chlamydia infection will reduce the disease activity in MS. The primary outcome measure will be reduction in new enhancing MS lesions on brain MRI. Forty patients will be entered into the trial. To be eligible, patients must have evidence of chlamydia infection in their spinal fluid and enhancing lesions on their pre-randomization MRI scans. Patients who meet these criteria will be randomized to either placebo or antibiotic therapy, and followed for 6 months on treatment.

ELIGIBILITY:
Patients with unequivocal diagnosis of multiple sclerosis and have evidence of C. pneumoniae infection in the cerebral spinal fluid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical School, Houston, Texas, United States